CLINICAL TRIAL: NCT02150590
Title: Patients With Chronic Obstructive Pulmonary Disease Staying at Altitude - Effect of Nocturnal Oxygen Therapy on Breathing and Sleep in
Brief Title: Patients With Chronic Obstructive Pulmonary Disease at Altitude - Effect of Nocturnal Oxygen on Breathing and Sleep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-0088V2A3B
Record Dates: First submitted 2014-05-18; First posted 2014-05-30 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: airway disease; bronchitis; emphysema; lung
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis; Emphysema | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxygen (Active Comparator): oxygen administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Interventions: Drug: Oxygen; Drug: sham oxygen (room air)
- Sham oxygen (Placebo Comparator): Sham oxygen (room air) administration via a nasal cannula at a rate of 3 L/min during nights spent at 2048 m
  Interventions: Drug: Oxygen; Drug: sham oxygen (room air)

INTERVENTIONS:
Drug: Oxygen — Nocturnal nasal oxygen during stay at 2048 m
Drug: sham oxygen (room air)
  Other Names: Nocturnal nasal room air during stay at 2048 m

SUMMARY:
The purpose of this study is to investigate the effect of nocturnal oxygen therapy during a stay at moderate altitude on breathing and sleep of patients with chronic obstructive lung disease.

DETAILED DESCRIPTION:
Patients with moderate to severe chronic obstructive pulmonary disease living below 800 m will be invited to participate in a randomized, cross-over field trial evaluating the hypothesis that nocturnal breathing and sleep during nights spent at moderate altitude are improved by oxygen therapy via a nasal cannula compared to room air (sham oxygen). Outcomes will be assessed at low altitude (Zurich, 490 m, baseline), and during 2 study periods of 2 nights each spent at moderate altitude (St. Moritz Salastrains, 2048 m) separated by a wash-out period of at least 2 weeks spent at low altitude (<800 m).

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease (COPD), GOLD grade 2-3
* residents at low altitude (<800 m)

Exclusion Criteria:

* unstable condition, COPD exacerbation
* mild (GOLD 1) or very severe COPD (GOLD 4)
* requirement for oxygen therapy at low altitude residence
* hypoventilation
* pulmonary hypertension
* more than mild or unstable cardiovascular disease
* use of drugs that affect respiratory center drive
* internal, neurologic or psychiatric disease that interfere with protocol compliance including current heavy smoking (>20 cigarettes per day), inability to perform 6 min walk test.
* previous intolerance to moderate altitude (<2600m).
* exposure to altitudes >1500m for >2 days within the last 4 weeks before the study.
* pregnant or nursing patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2014-10-31 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | Approximately 8 hours (during the first night at 2048 m)
  Difference in mean nocturnal oxygen saturation between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Apnea/hypopnea index measured by polysomnography | Approximately 8 hours (during the first night at 2048 m)
  Difference in apnea/hypopnea index between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.

SECONDARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | Approximately 8 hours (during the second night at 2048 m)
  Difference in mean nocturnal oxygen saturation between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Apnea/hypopnea index measured by polygraphy | Approximately 8 hours (during the second night at 2048 m)
  Difference in apnea/hypopnea index between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Subjective sleep quality visual analog scale score | Approximately 8 hours (during the first night at 2048 m)
  Difference in subjective sleep quality visual analog scale scores between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Psychomotor vigilance test reaction time | Approximately at 10 a.m. on the second day at 2048 m
  Difference in subjective sleep quality between visual analog scale measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.
Severe hypoxemia | Approximately 72 hours (day 1 to 3 at 2048 m)
  Number of participants in whom arterial oxygen saturation measured by pulse oximetry is less than 75% for more than 30 min during the oxygen and sham oxygen treatment periods at 2028 m.
Subjective sleep quality visual analog scale score | Approximately 8 hours (during the second night at 2048 m)
  Difference in subjective sleep quality visual analog scale scores between measurements at 2048 m (altitude) and 490 m (baseline); and between the oxygen and sham oxygen treatment periods at 2048 m.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland

REFERENCES:
- [Derived] Gutweniger S, Latshang TD, Aeschbacher SS, Huber F, Flueck D, Lichtblau M, Ulrich S, Hasler ED, Scheiwiller PM, Ulrich S, Bloch KE, Furian M. Effect of nocturnal oxygen therapy on exercise performance of COPD patients at 2048 m: data from a randomized clinical trial. Sci Rep. 2021 Oct 13;11(1):20355. doi: 10.1038/s41598-021-98395-w. PMID 34645842
- [Derived] Lichtblau M, Latshang TD, Aeschbacher SS, Huber F, Scheiwiller PM, Ulrich S, Schneider SR, Hasler ED, Furian M, Bloch KE, Saxer S, Ulrich S. Effect of Nocturnal Oxygen Therapy on Daytime Pulmonary Hemodynamics in Patients With Chronic Obstructive Pulmonary Disease Traveling to Altitude: A Randomized Controlled Trial. Front Physiol. 2021 Jul 7;12:689863. doi: 10.3389/fphys.2021.689863. eCollection 2021. PMID 34305642
- [Derived] Tan L, Latshang TD, Aeschbacher SS, Huber F, Flueck D, Lichtblau M, Ulrich S, Hasler ED, Scheiwiller PM, Ulrich S, Bloch KE, Furian M. Effect of Nocturnal Oxygen Therapy on Nocturnal Hypoxemia and Sleep Apnea Among Patients With Chronic Obstructive Pulmonary Disease Traveling to 2048 Meters: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207940. doi: 10.1001/jamanetworkopen.2020.7940. PMID 32568400